CLINICAL TRIAL: NCT06062550
Title: Efficacy of Different Dose Esketamine and Dexmedetomidine Combination for Supplemental Analgesia After Scoliosis Correction Surgery: A Randomized, Double-blind Trial
Brief Title: Different Dose Esketamine and Dexmedetomidine Combination for Supplemental Analgesia After Scoliosis Correction Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023-351
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Scoliosis Correction; Esketamine; Dexmedetomidine; Postoperative Analgesia; Chronic Postsurgical Pain
Keywords: Scoliosis Correction; Esketamine; Dexmedetomidine; Postoperative Analgesia; Chronic Postsurgical Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-dose group (Active Comparator): Patient-controlled analgesia is established with esketamine 50 mg, dexmedetomidine 200 microgram, and sufentanil 4 microgram/kg (maximum 250 microgram), diluted with normal saline to 200 ml, and programmed to administer 2-ml boluses with a lockout interval of 8 minutes and a background infusion rate at 1 ml/h.
  Interventions: Drug: Esketamine
- Medium-dose group (Experimental): Patient-controlled analgesia is established with esketamine 100 mg, dexmedetomidine 200 microgram, and sufentanil 4 microgram/kg (maximum 250 microgram), diluted with normal saline to 200 ml, and programmed to administer 2-ml boluses with a lockout interval of 8 minutes and a background infusion rate at 1 ml/h.
  Interventions: Drug: Esketamine
- High-dose group (Experimental): Patient-controlled analgesia is established with esketamine 150 mg, dexmedetomidine 200 microgram, and sufentanil 4 microgram/kg (maximum 250 microgram), diluted with normal saline to 200 ml, and programmed to administer 2-ml boluses with a lockout interval of 8 minutes and a background infusion rate at 1 ml/h.
  Interventions: Drug: Esketamine

INTERVENTIONS:
Drug: Esketamine — Different doses of esketamine in the esketamine-dexmedetomidine combination as a supplement to sufentanil for postoperative intravenous analgesia.

SUMMARY:
Scoliosis correction surgery is associated with severe pain. Patients after scoliosis correction surgery usually require high dose opioids and long duration analgesia, which may increase side effects and drug tolerance. In a recent trial, mini-dose esketamine and dexmedetomidine combination as a supplement to sufentanil significantly improved analgesia and subjective sleep quality after spinal correction surgery without increasing adverse events; however, the proportion of patients with moderate-to-severe pain remained high. The authors speculate that increasing esketamine dose in the combination may further improve analgesic effects.

DETAILED DESCRIPTION:
Spinal surgery is associated with severe pain, with a median pain score of 7 (interquartile range, 4 to 8) on the first postoperative day, and requires long duration analgesia. The total dose of opioids required for postoperative analgesia is about 2-4 times that for other surgeries. However, despite high dose opioids, the analgesic effects remain unsatisfied. In a recent trial of 200 patients following scoliosis correction surgery, the proportion with moderate-to-severe pain in patients given routine analgesia was 84.6%. Severe acute pain is an important risk factor of chronic postsurgical pain and is associated with an increased risk of long-term opioid use.

Ketamine is a non-competitive N-methyl-D-aspartate receptor antagonist. Low-dose ketamine infusion is recommended for postoperative analgesia but may cause neuropsychiatric side effects. Esketamine is the S-enantiomer of racemic ketamine with approximately twice as potent as racemic ketamine in analgesia and less likely to produce side effects. Dexmedetomidine is a highly selective α2 receptor agonist and has anxiolytic, sedative, analgesic effects. When used as a supplement to opioid analgesia, dexmedetomidine improves analgesia and sleep quality but may produce sedation.

In a recent trial, mini-dose esketamine-dexmedetomidine combination as a supplement to sufentanil significantly improved analgesia and subjective sleep quality after scoliosis correction surgery; no significant adverse reactions were observed. However, the proportion of moderate-to-severe pain remained high (65.7%) in these patients, so further improvement is needed. The authors speculate that increasing esketamine dose in the esketamine-dexmedetomidine combination may further improve the analgesia. This study aims to explore the effects of different dose esketamine in the combination on acute and chronic pain in patients following spinal deformity surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years and body weight ≥40 kg;
* Scheduled to undergo scoliosis correction with pedicle screw fixation;
* Required patient-controlled intravenous analgesia after surgery.

Exclusion Criteria:

* Preoperative sick sinus syndrome, severe sinus bradycardia (heart rate <50 beats/min), atrioventricular block grade II or above without pacemaker; or comorbid with congenital heart disease, arrhythmia, or other serious cardiovascular diseases with a cardiac function grade ≥III;
* Patients with moderate and severe obstructive sleep apnea diagnosed preoperatively or according to the STOP-Bang score；
* History of hyperthyroidism and pheochromocytoma;
* History of schizophrenia, epilepsy, myasthenia gravis, or delirium;
* Severe liver dysfunction (child Pugh grade C), severe renal dysfunction (preoperative dialysis), or American Society of Anesthesiologists grade ≥IV;
* Barrier in communication;
* Other conditions that are considered unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Pain intensity with movement and opioid consumption within 72 hours. | Within 72 hours after surgery
  A comprehensive index of pain intensity and opioid consumption is calculated. The range of the index is -200% to +200%; values above 0 indicate increased summed area under curve (AUC) and opioid consumption (OC) compared to the all patients.

SECONDARY OUTCOMES:
Proportion of patients with moderate to severe pain within 72 hours. | Up to 72 hours after surgery.
  Pain intensity is evaluated with the Numeric Rating Scale (NRS, an 11-point scale where 0 = no pain and 10 = the worst pain) twice daily (8:00-10:00 and 18:00-20:00) at rest and with movement. Moderate to severe pain is defined as any NRS pain score of 4 or higher.
The highest NRS pain score within 72 hours after surgery. | Up to 72 hours after surgery.
  Pain intensity is evaluated with the Numeric Rating Scale (NRS, an 11-point scale where 0 = no pain and 10 = the worst pain) twice daily (8:00-10:00 and 18:00-20:00) at rest and with movement.
Area under curve of NRS pain score within 72 hours after surgery. | Up to 72 hours after surgery
  Pain intensity is evaluated with the Numeric Rating Scale (NRS, an 11-point scale where 0 = no pain and 10 = the worst pain) twice daily (8:00-10:00 and 18:00-20:00) at rest and with movement.
Cumulative opioid consumption within 72 hours after surgery. | Up to 72 hours after surgery
  Cumulative opioid consumption within 72 hours after surgery.
Requirement of supplement analgesia within 72 hours. | Up to 72 hours after surgery
  Requirement of supplement analgesia within 72 hours.
Pain intensity at rest and opioid consumption within 72 hours. | Within 72 hours after surgery.
  A comprehensive index of pain intensity and opioid consumption is calculated. The range of the index is -200% to +200%; values above 0 indicate increased summed AUC and OC compared to the all patients.
Subjective sleep quality during the first 5 postoperative days. | Up to the 5th day after surgery.
  Subjective sleep quality is evaluated with the Numeric Rating Scale (NRS, an 11-point scale where 0 = the best sleep and 10 = no sleep at all) once daily (8:00-10:00).
Number of days requiring analgesics within 30 days after surgery. | Up to 30 days after surgery.
  Number of days requiring analgesics within 30 days after surgery.

OTHER OUTCOMES:
Agitation and sedation score at various timepoints after surgery. | Up to the 5th day after surgery.
  Agitation and sedation score is evaluated with the Richmond Agitation and Sedation Scale (RASS, with scores ranging from -5 [unarousable] to +4 [combative] and 0 indicates alert and calm) twice daily (8:00-10:00 and 18:00-20:00).
Incidence of postoperative delirium within the first 5 days. | Up to the 5th day after surgery.
  Delirium is assessed with the Three-dimensional Confusion Assessment Method (3D-CAM) twice daily (8:00-10:00 and 18:00-20:00).
Depression severity at 7 days after surgery. | At the 7th day after surgery.
  Depression is assessed with the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 includes 9-item requiring responses of 0 (not at all) to 3 (nearly every day) to assess the occurrence of depressive symptoms over the last two weeks. It has 8 items on depressive symptoms and 1 focused on suicidal ideation. Total scores range from 0 to 27, with higher score indicating more severe symptoms.
Length of stay in hospital after surgery. | Up to 30 days after surgery.
  Length of stay in hospital after surgery.
Incidence of postoperative complications within 30 days | Up to 30 days after surgery.
  Postoperative complications are defined as new-onset medical conditions that were deemed harmful and required therapeutic intervention (i.e., grade II or higher on the Clavien-Dindo classification).

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD,PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Beijing University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Hussain A, Erdek M. Interventional pain management for failed back surgery syndrome. Pain Pract. 2014 Jan;14(1):64-78. doi: 10.1111/papr.12035. Epub 2013 Feb 3. PMID 23374545
- [Background] Wylde V, Dennis J, Beswick AD, Bruce J, Eccleston C, Howells N, Peters TJ, Gooberman-Hill R. Systematic review of management of chronic pain after surgery. Br J Surg. 2017 Sep;104(10):1293-1306. doi: 10.1002/bjs.10601. Epub 2017 Jul 6. PMID 28681962
- [Background] Dunn LK, Yerra S, Fang S, Hanak MF, Leibowitz MK, Tsang S, Durieux ME, Nemergut EC, Naik BI. Incidence and Risk Factors for Chronic Postoperative Opioid Use After Major Spine Surgery: A Cross-Sectional Study With Longitudinal Outcome. Anesth Analg. 2018 Jul;127(1):247-254. doi: 10.1213/ANE.0000000000003338. PMID 29570151
- [Background] Leider HL, Dhaliwal J, Davis EJ, Kulakodlu M, Buikema AR. Healthcare costs and nonadherence among chronic opioid users. Am J Manag Care. 2011 Jan;17(1):32-40. PMID 21348566
- [Background] Schwenk ES, Viscusi ER, Buvanendran A, Hurley RW, Wasan AD, Narouze S, Bhatia A, Davis FN, Hooten WM, Cohen SP. Consensus Guidelines on the Use of Intravenous Ketamine Infusions for Acute Pain Management From the American Society of Regional Anesthesia and Pain Medicine, the American Academy of Pain Medicine, and the American Society of Anesthesiologists. Reg Anesth Pain Med. 2018 Jul;43(5):456-466. doi: 10.1097/AAP.0000000000000806. PMID 29870457
- [Background] Cohen SP, Bhatia A, Buvanendran A, Schwenk ES, Wasan AD, Hurley RW, Viscusi ER, Narouze S, Davis FN, Ritchie EC, Lubenow TR, Hooten WM. Consensus Guidelines on the Use of Intravenous Ketamine Infusions for Chronic Pain From the American Society of Regional Anesthesia and Pain Medicine, the American Academy of Pain Medicine, and the American Society of Anesthesiologists. Reg Anesth Pain Med. 2018 Jul;43(5):521-546. doi: 10.1097/AAP.0000000000000808. PMID 29870458
- [Background] Molero P, Ramos-Quiroga JA, Martin-Santos R, Calvo-Sanchez E, Gutierrez-Rojas L, Meana JJ. Antidepressant Efficacy and Tolerability of Ketamine and Esketamine: A Critical Review. CNS Drugs. 2018 May;32(5):411-420. doi: 10.1007/s40263-018-0519-3. PMID 29736744
- [Background] Canuso CM, Singh JB, Fedgchin M, Alphs L, Lane R, Lim P, Pinter C, Hough D, Sanacora G, Manji H, Drevets WC. Efficacy and Safety of Intranasal Esketamine for the Rapid Reduction of Symptoms of Depression and Suicidality in Patients at Imminent Risk for Suicide: Results of a Double-Blind, Randomized, Placebo-Controlled Study. Am J Psychiatry. 2018 Jul 1;175(7):620-630. doi: 10.1176/appi.ajp.2018.17060720. Epub 2018 Apr 16. PMID 29656663
- [Background] Segmiller F, Ruther T, Linhardt A, Padberg F, Berger M, Pogarell O, Moller HJ, Kohler C, Schule C. Repeated S-ketamine infusions in therapy resistant depression: a case series. J Clin Pharmacol. 2013 Sep;53(9):996-8. doi: 10.1002/jcph.122. Epub 2013 Jul 24. No abstract available. PMID 23893490
- [Background] Persson J, Hasselstrom J, Maurset A, Oye I, Svensson JO, Almqvist O, Scheinin H, Gustafsson LL, Almqvist O. Pharmacokinetics and non-analgesic effects of S- and R-ketamines in healthy volunteers with normal and reduced metabolic capacity. Eur J Clin Pharmacol. 2002 Feb;57(12):869-75. doi: 10.1007/s002280100353. PMID 11936706
- [Background] Loftus RW, Yeager MP, Clark JA, Brown JR, Abdu WA, Sengupta DK, Beach ML. Intraoperative ketamine reduces perioperative opiate consumption in opiate-dependent patients with chronic back pain undergoing back surgery. Anesthesiology. 2010 Sep;113(3):639-46. doi: 10.1097/ALN.0b013e3181e90914. PMID 20693876
- [Background] Nielsen RV, Fomsgaard JS, Siegel H, Martusevicius R, Nikolajsen L, Dahl JB, Mathiesen O. Intraoperative ketamine reduces immediate postoperative opioid consumption after spinal fusion surgery in chronic pain patients with opioid dependency: a randomized, blinded trial. Pain. 2017 Mar;158(3):463-470. doi: 10.1097/j.pain.0000000000000782. PMID 28067693
- [Background] Nielsen RV, Fomsgaard JS, Nikolajsen L, Dahl JB, Mathiesen O. Intraoperative S-ketamine for the reduction of opioid consumption and pain one year after spine surgery: A randomized clinical trial of opioid-dependent patients. Eur J Pain. 2019 Mar;23(3):455-460. doi: 10.1002/ejp.1317. Epub 2018 Oct 14. PMID 30246357
- [Background] Nielsen RV. Adjuvant analgesics for spine surgery. Dan Med J. 2018 Mar;65(3):B5468. PMID 29510816
- [Background] Carley ME, Chaparro LE, Choiniere M, Kehlet H, Moore RA, Van Den Kerkhof E, Gilron I. Pharmacotherapy for the Prevention of Chronic Pain after Surgery in Adults: An Updated Systematic Review and Meta-analysis. Anesthesiology. 2021 Aug 1;135(2):304-325. doi: 10.1097/ALN.0000000000003837. PMID 34237128
- [Background] Stone LS, MacMillan LB, Kitto KF, Limbird LE, Wilcox GL. The alpha2a adrenergic receptor subtype mediates spinal analgesia evoked by alpha2 agonists and is necessary for spinal adrenergic-opioid synergy. J Neurosci. 1997 Sep 15;17(18):7157-65. doi: 10.1523/JNEUROSCI.17-18-07157.1997. PMID 9278550
- [Background] Peng K, Zhang J, Meng XW, Liu HY, Ji FH. Optimization of Postoperative Intravenous Patient-Controlled Analgesia with Opioid-Dexmedetomidine Combinations: An Updated Meta-Analysis with Trial Sequential Analysis of Randomized Controlled Trials. Pain Physician. 2017 Nov;20(7):569-596. PMID 29149140
- [Background] Wu XH, Cui F, Zhang C, Meng ZT, Wang DX, Ma J, Wang GF, Zhu SN, Ma D. Low-dose Dexmedetomidine Improves Sleep Quality Pattern in Elderly Patients after Noncardiac Surgery in the Intensive Care Unit: A Pilot Randomized Controlled Trial. Anesthesiology. 2016 Nov;125(5):979-991. doi: 10.1097/ALN.0000000000001325. PMID 27571256
- [Background] Bornemann-Cimenti H, Wejbora M, Michaeli K, Edler A, Sandner-Kiesling A. The effects of minimal-dose versus low-dose S-ketamine on opioid consumption, hyperalgesia, and postoperative delirium: a triple-blinded, randomized, active- and placebo-controlled clinical trial. Minerva Anestesiol. 2016 Oct;82(10):1069-1076. Epub 2016 Jun 21. PMID 27327855
- [Background] Hu ZC, Xu G, Zhang XW, Ma K, Jin JJ, Li PS. [Meta-analysis of the effects of dexmedetomidine combined with ketamine during dressing changes in burn patients]. Zhonghua Shao Shang Za Zhi. 2020 Jun 20;36(6):458-464. doi: 10.3760/cma.j.cn501120-20190327-00145. Chinese. PMID 32594705
- [Background] Lee KH, Lee SJ, Park JH, Kim SH, Lee H, Oh DS, Kim YH, Park YH, Kim H, Lee SE. Analgesia for spinal anesthesia positioning in elderly patients with proximal femoral fractures: Dexmedetomidine-ketamine versus dexmedetomidine-fentanyl. Medicine (Baltimore). 2020 May;99(20):e20001. doi: 10.1097/MD.0000000000020001. PMID 32443302
- [Background] Brinck ECV, Virtanen T, Makela S, Soini V, Hynninen VV, Mulo J, Savolainen U, Rantakokko J, Maisniemi K, Liukas A, Olkkola KT, Kontinen V, Tarkkila P, Peltoniemi M, Saari TI. S-ketamine in patient-controlled analgesia reduces opioid consumption in a dose-dependent manner after major lumbar fusion surgery: A randomized, double-blind, placebo-controlled clinical trial. PLoS One. 2021 Jun 7;16(6):e0252626. doi: 10.1371/journal.pone.0252626. eCollection 2021. PMID 34097713
- [Background] Nagappa M, Wong J, Singh M, Wong DT, Chung F. An update on the various practical applications of the STOP-Bang questionnaire in anesthesia, surgery, and perioperative medicine. Curr Opin Anaesthesiol. 2017 Feb;30(1):118-125. doi: 10.1097/ACO.0000000000000426. PMID 27898430
- [Background] Andersen LPK, Gogenur I, Torup H, Rosenberg J, Werner MU. Assessment of Postoperative Analgesic Drug Efficacy: Method of Data Analysis Is Critical. Anesth Analg. 2017 Sep;125(3):1008-1013. doi: 10.1213/ANE.0000000000002007. PMID 28632527
- [Background] Cheung KM, Senkoylu A, Alanay A, Genc Y, Lau S, Luk KD. Reliability and concurrent validity of the adapted Chinese version of Scoliosis Research Society-22 (SRS-22) questionnaire. Spine (Phila Pa 1976). 2007 May 1;32(10):1141-5. doi: 10.1097/01.brs.0000261562.48888.e3. PMID 17471100
- [Background] Li M, Wang CF, Gu SX, He SS, Zhu XD, Zhao YC, Zhang JT. Adapted simplified Chinese (mainland) version of Scoliosis Research Society-22 questionnaire. Spine (Phila Pa 1976). 2009 May 20;34(12):1321-4. doi: 10.1097/BRS.0b013e31819812b7. PMID 19455008
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912